CLINICAL TRIAL: NCT01286246
Title: Pilot Randomized Controlled Trial of Vaginal Progesterone to Prevent Preterm Birth in Women With Threatened Preterm Labor
Brief Title: Randomized Controlled Trial of Vaginal Progesterone in Women With Threatened Preterm Labor
Acronym: PROTO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Trial investigators were unable to recruit the estimated sample
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Sue Ross, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21492
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Obstetric Labor, Premature
Keywords: Progesterone; Randomized controlled trial
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Utrogestan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaginal progesterone (Experimental)
  Interventions: Drug: Vaginal progesterone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vaginal progesterone — Capsules of 200mg micronised progesterone suspended in sunflower oil. One capsule inserted vaginally per day from time of randomisation to gestational age 35(+6)weeks or delivery (if sooner).
  Other Names: Utrogestan
  Arms: Vaginal progesterone
Drug: Placebo — Capsules of placebo (sunflower oil). One capsule inserted vaginally per day from time of randomisation to gestational age 35(+6)weeks or delivery (if sooner).
  Arms: Placebo

SUMMARY:
Prematurity remains the most important single factor in perinatal morbidity and mortality. Unfortunately, the rate of premature delivery is increasing in Canada and is especially high in Alberta with 7.5% of pregnancies ending before 37 weeks gestation. Despite years of research into the causes of spontaneous preterm labor, few effective treatments have been identified. Progesterone is one candidate treatment. The purpose of this study is to investigate whether progesterone can prolong pregnancy in women who have symptoms of preterm labor.

Pregnant women who have symptoms of premature labor will be invited to take part in the study if they are between 22 to 24 weeks pregnant. If they agree to join the study, they will be randomly allocated to either take progesterone 200mg each day via the vagina until 36 weeks, or to take a placebo preparation. Neither the women nor their clinician will know which group they are in.

Women and their babies will be followed until 28 days after the birth, to find out about the length of the pregnancy, any adverse events that might occur (none have been reported in previous trials), and to look at whether women have taken the treatment.

When the study is complete, the results for the progesterone group will be compared to the placebo group. If progesterone is found to be useful in helping to prolong pregnancy, then this will be a possible treatment to help mothers in the future.

ELIGIBILITY:
Inclusion Criteria:

* Women with symptomatic premature contractions successfully arrested for at least 12 hours with tocolytics.
* Women with symptoms suggestive of early preterm labor whose contractions resolve without tocolysis but are fetal fibronectin positive.
* Gestational age 23(+0)-32(+6) weeks.
* Consent to taking part in the study.

Exclusion Criteria:

* Placenta previa
* Preterm premature rupture of membranes at presentation
* Pre-existing hypertension will be excluded in order to reduce the likelihood of iatrogenic preterm delivery within the study women
* Known major fetal anomaly detected on ultrasound
* Multiple pregnancy
* Maternal seizure disorder
* Active or history of thromboembolic disease
* Maternal liver disease
* Known or suspected breast malignancy or pathology
* Known or suspected progesterone-dependent neoplasia
* Plans to move to another city during pregnancy
* Previous participation in a progesterone trial during this pregnancy
* Known sensitivity to progesterone

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2011-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Gestational age at birth | At birth
  Gestational age at birth calculated from gestational age at pre-randomization baseline

SECONDARY OUTCOMES:
Proportion of women who have preterm birth <35 weeks | At birth
Proportion of women who have a preterm birth at <37 weeks | At birth
Maternal hospital length of stay (days) | Days from date of admission to date of discharge
Proportion of women who have hospital admission for premature labor | After birth
Maternal compliance with treatment | At time of birth
  Diary self-report of treatment use
Neonatal hospital length of stay (days) | Days from birth to discharge from hospital
Neonatal morbidity | Up to 28 days after birth
  Respiratory distress syndrome (type 1), intraventricular hemorrhage, chronic lung disease, periventricular leukomalacia,necrotising eneterocolitis, retinopathy of prematurity
Number of days of assisted ventilation (neonate) | Up to 28 days after birth
Number of days of supplemental oxygen (for neonate) | Up to 28 days after birth
Birth weight (grams) | At time of birth
Neonatal survival to discharge home (yes/no) | During 28 days after birth
Adverse events (maternal or neonate) | Up to 28 days after birth

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Wood, MD, MSc, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada